CLINICAL TRIAL: NCT01888159
Title: Salpingectomy vs Tubal Sterilisation in Low Risk for Ovarian Cancer Women and Its Effect on Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Leonidas Magarakis, MD, Karlstad Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEvsTSinAMH
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sterilization, Tubal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tubal Sterilization with bipolar (Active Comparator): Salpingectomy vs Tubal Sterilisation
  Interventions: Procedure: Tubal sterilization with bipolar energy
- Bilateral Salpingectomy (Active Comparator): Salpingectomy vs Tubal Sterilisation
  Interventions: Procedure: Bilateral Salpingectomy

INTERVENTIONS:
Procedure: Bilateral Salpingectomy
  Arms: Bilateral Salpingectomy
Procedure: Tubal sterilization with bipolar energy
  Arms: Tubal Sterilization with bipolar

SUMMARY:
Randomised study to investigate if salpingectomies done to women wishing tubal sterilisation has an effect on ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking for tubal sterilisation

Exclusion Criteria:

* women older than 45
* family history of ovarian cancer
* presence of menopausal symptoms
* irregular cycles
* Hormone Replacement Therapy or hormone contraceptions the last 3 months
* history of previous ovarian or uterine surgeries
* imaging suggesting an ovarian cyst or other adnexal pathology during investigation
* previous salpingectomy

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian hormone (AMH)and Follicle Stimulation Hormone (FSH) | 3 months

SECONDARY OUTCOMES:
Anti-Mullerian hormone (AMH) | 1 year
Operative time | Postoperatively
Complications | 3 months

OTHER OUTCOMES:
Follicle Stimulation Hormone (FSH) | 3 months
Follicle Stimulation Hormone (FSH) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Karlstad, Värmaland, Sweden